CLINICAL TRIAL: NCT04049617
Title: A Phase 1b/2 Dose Escalation/Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of GS-4224 in Subjects With Advanced Solid Tumors
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Evixapodlin (Formerly GS-4224) in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Gilead decision to terminate
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-494-5484; 2019-004605-27 (EudraCT Number)
Record Dates: First submitted 2019-07-31; First posted 2019-08-08 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1: Evixapodlin 400 mg (Phase 1) (Experimental): Participants will receive Evixapodlin 400 mg once daily for 21 days of each cycle.
  Interventions: Drug: Evixapodlin
- Cohort 2: Evixapodlin 700 mg (Phase 1) (Experimental): Participants will receive Evixapodlin 700 mg once daily for 21 days of each cycle.
  Interventions: Drug: Evixapodlin
- Cohort 3: Evixapodlin 1000 mg (Phase 1) (Experimental): Participants will receive Evixapodlin 1000 mg once daily for 21 days of each cycle.
  Interventions: Drug: Evixapodlin
- Cohort 4: Evixapodlin 1500 mg (Phase 1) (Experimental): Participants will receive Evixapodlin 1500 mg once daily for 21 days of each cycle.
  Interventions: Drug: Evixapodlin
- Cohort 5: Evixapodlin 1000 mg (Phase 1) (Experimental): Participants are planned to receive Evixapodlin 1000 mg twice daily (BID) for 21 days of each cycle.
  Interventions: Drug: Evixapodlin
- Cohort 1 Substudy: Evixapodlin 400 mg (Phase 1) (Experimental): Participants will receive Evixapodlin 400 mg once daily for 21 days of each cycle.
  Interventions: Drug: Evixapodlin
- Cohort 2 Substudy: Evixapodlin 700 mg (Phase 1) (Experimental): Participants are planned to receive Evixapodlin 700 mg once daily for 21 days of each cycle.
  Interventions: Drug: Evixapodlin
- Cohort 3 Substudy: Evixapodlin 1000 mg (Phase 1) (Experimental): Participants will receive Evixapodlin 1000 mg once daily for 21 days of each cycle.
  Interventions: Drug: Evixapodlin
- Dose Expansion (Phase 2) (Experimental): Dose expansion is planned to begin when the recommended Phase 2 dose (RP2D) will be determined.
  Interventions: Drug: Evixapodlin

INTERVENTIONS:
Drug: Evixapodlin — Tablets administered orally.
  Other Names: GS-4224

SUMMARY:
The primary objectives of this study are to characterize the safety and tolerability of evixapodlin (formerly GS-4224) and to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of evixapodlin in participants with advanced solid tumors.

DETAILED DESCRIPTION:
This was a planned Phase 1/2 study. However, Phase 2 was not conducted because the study was closed due to sponsor decision prior to opening the dose expansion cohort and hence, RP2D analysis was not performed.

ELIGIBILITY:
Key Inclusion Criteria:

* Dose Escalation Cohorts: Histologically or cytologically confirmed advanced malignant solid tumor that is refractory to or intolerant of all standard therapy or for which no standard therapy is available.
* Dose Expansion and 1000 mg twice a day (BID) Dose Escalation Cohorts: Individuals must have available sufficient and adequate formalin fixed tumor sample preferably from a biopsy of a tumor lesion obtained either at the time of or after the diagnosis of advanced disease has been made and from a site not previously irradiated. Alternatively, individuals must agree to have a biopsy taken prior to entering the study to provide adequate tissue. For the 1000 mg BID dose escalation cohort, individuals with melanoma, Merkel cell, microsatellite instability-high (MSI-H) cancers, and classical Hodgkin lymphoma (cHL) are not required to have archival or fresh biopsy tissue.
* Dose Escalation Biopsy Substudy and 1000 mg BID Dose Escalation Cohorts: Documented ligand 1 of programmed cell death protein 1 (PD-L1) expression in the tumor (tumor proportion score (TPS) ≥ 10% or combined positive score (CPS) ≥ 10). In the 1000 mg BID Cohort, PD-L1 expression will not be required for Merkel cell, melanoma, MSI-H cancers, and cHL.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Adequate organ function.

Key Exclusion Criteria:

* History or evidence of clinically significant disorder, condition, or disease that, in the opinion of the Investigator or Medical Monitor would pose a risk to individual safety or interfere with the study evaluations, procedures, or completion.
* Dose Escalation Cohorts: History of ≥ Grade 3 Adverse Events (AEs) during prior treatment with an immune checkpoint inhibitor, or history of discontinuation of treatment with an immune checkpoint inhibitor due to AEs.
* Dose Escalation 1000 mg BID and Dose Expansion Cohort: Prior treatment with an immune checkpoint inhibitor (anti-PD-1, anti-PD-L1, or anti- ligand 2 of programmed cell death protein 1 (PD-L2) antibodies).
* History of autoimmune disease (for example, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (3):
  - California Care Associates for Research and Excellence Inc, Encinitas, California
  - NEXT Oncology, San Antonio, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Clinical Studies Trust, LLC, Christchurch
  - Auckland Clinical Studies Ltd, Grafton, Auckland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Odegard JM, Othman AA, Lin KW, Wang AY, Nazareno J, Yoon OK, Ling J, Lad L, Dunbar PR, Thai D, Ang E, Waldron N, Deva S. Oral PD-L1 inhibitor GS-4224 selectively engages PD-L1 high cells and elicits pharmacodynamic responses in patients with advanced solid tumors. J Immunother Cancer. 2024 Apr 11;12(4):e008547. doi: 10.1136/jitc-2023-008547. PMID 38604815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in New Zealand and the United States. The first participant was screened on 26 August 2019. The last study visit occurred on 30 March 2021.
Pre-assignment Details: 29 participants were screened. The participants took part in the Phase 1 (Dose Escalation) of the study only. No participants were enrolled in the Phase 1 Cohort 5 and Cohort 2 substudy and the study was terminated due to sponsor decision before the planned Dose Expansion Phase 2 started.
Groups:
- Cohort 1: Evixapodlin 400 mg (Phase 1): Participants received evixapodlin 400 mg once daily for 21 days of each cycle (observed maximum duration was approximately 21 weeks).
- Cohort 2: Evixapodlin 700 mg (Phase 1): Participants received evixapodlin 700 mg once daily for 21 days of each cycle (observed maximum duration was approximately 10 weeks).
- Cohort 3: Evixapodlin 1000 mg (Phase 1): Participants received evixapodlin 1000 mg once daily for 21 days of each cycle (observed maximum duration was approximately 39 weeks).
- Cohort 4: Evixapodlin 1500 mg (Phase 1): Participants received evixapodlin 1500 mg once daily for 21 days of each cycle (observed maximum duration was approximately 19 weeks).
- Cohort 1 Substudy: Evixapodlin 400 mg (Phase 1): Participants received evixapodlin 400 mg once daily for 21 days of each cycle (observed maximum duration was approximately 39 weeks).
- Cohort 3 Substudy: Evixapodlin 1000 mg (Phase 1): Participants received evixapodlin 1000 mg once daily for 21 days of each cycle (observed maximum duration was approximately 10 weeks).
Period: Overall Study
Arm/Group | Cohort 1: Evixapodlin 400 mg (Phase 1) | Cohort 2: Evixapodlin 700 mg (Phase 1) | Cohort 3: Evixapodlin 1000 mg (Phase 1) | Cohort 4: Evixapodlin 1500 mg (Phase 1) | Cohort 1 Substudy: Evixapodlin 400 mg (Phase 1) | Cohort 3 Substudy: Evixapodlin 1000 mg (Phase 1)
Started | 3 | 3 | 6 | 3 | 2 | 1
Completed | 3 | 3 | 5 | 1 | 2 | 0
Not Completed | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included data from all participants who received at least 1 dose of study treatment, with treatment assignments designated according to the actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Evixapodlin 400 mg (Phase 1) | Cohort 2: Evixapodlin 700 mg (Phase 1) | Cohort 3: Evixapodlin 1000 mg (Phase 1) | Cohort 4: Evixapodlin 1500 mg (Phase 1) | Cohort 1 Substudy: Evixapodlin 400 mg (Phase 1) | Cohort 3 Substudy: Evixapodlin 1000 mg (Phase 1) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 2 | 1 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (28.29) | 65.3 (15.53) | 61.2 (5.67) | 70.0 (11.53) | 64.0 (12.73) | 42.0 (NA) — Due to less number of participants, standard deviation was not estimable. | 61.6 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 0 | 0 | 0 | 3
  Male | 2 | 3 | 4 | 3 | 2 | 1 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 2 | 5 | 2 | 2 | 0 | 12
  United States | 2 | 1 | 1 | 1 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicities (DLTs) During the Dose Escalation Phase
Description: A DLT was any toxicity defined as follows excluding toxicities clearly related to disease progression or disease-related processes occurring during the DLT assessment window (Day 1 through Day 21):
  * Grade ≥ 4 neutropenia
  * Grade ≥ 3 neutropenia with fever
  * Grade ≥ 3 thrombocytopenia
  * Grade ≥ 2 bleeding
  * Grade ≥ 3 anemia
  * Grade ≥ 3 or higher non-hematologic toxicity (excluding Grade 3 nausea or emesis or Grade 3 diarrhea)
  * Grade ≥ 2 non-hematologic treatment-emergent adverse event that in the opinion of the investigator is of potential clinical significance
  * Treatment interruption of ≥ 7 days due to unresolved toxicity
  * Any toxicity event that precludes further administration of evixapodlin
  * Any Grade 3 or Grade 4 elevation in aspartate aminotransferase (AST) or alanine aminotransferase (ALT) associated with a Grade 2 elevation in bilirubin lasting ≥ 7 days
  * An immune-related adverse event (irAE) for which immunotherapy should be permanently discontinued
Time Frame: Day 1 through Day 21
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Evixapodlin 400 mg (Phase 1) | Cohort 2: Evixapodlin 700 mg (Phase 1) | Cohort 3: Evixapodlin 1000 mg (Phase 1) | Cohort 4: Evixapodlin 1500 mg (Phase 1) | Cohort 1 Substudy: Evixapodlin 400 mg (Phase 1) | Cohort 3 Substudy: Evixapodlin 1000 mg (Phase 1)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 2 | 1
Participants | 0 | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Evixapodlin During the Dose Escalation Phase
Description: AUCtau was defined as area under the concentration-time curve from time zero to the end of the dosing interval.
Time Frame: Intensive PK: Predose, 0.5, 1, 1.5, 2.5, 4, 6, 24 hours (h) postdose (400-1500 once daily [QD] mg cohorts) on Cycle (C) 1 Day (D) 1 & D15
Population: PK Analysis Set included participants in the Safety Analysis Set who had received the study drug and have at least 1 sample with detectable drug concentration. Data for Cohort 1 included participants from Cohort 1 and Substudy Cohort 1. PK data were not collected for Cohort 3 Substudy group due to discontinuation of the development program.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Cohort 4: Evixapodlin1500 mg (Phase 1): Participants received evixapodlin 1500 mg once daily for 21 days of each cycle (observed maximum duration was approximately 19 weeks).
Arm/Group | Cohort 1: Evixapodlin 400 mg (Phase 1) | Cohort 2: Evixapodlin 700 mg (Phase 1) | Cohort 3: Evixapodlin 1000 mg (Phase 1) | Cohort 4: Evixapodlin1500 mg (Phase 1)
Number analyzed (Participants) | 5 | 3 | 6 | 3
h*ng/mL
  C1D1 | 6543.1 (1783.07) | 8703.8 (3717.93) | 12241.8 (2793.17) | 19132.6 (596.64)
  C1D15 | 9269.8 (2693.53) | 13508.4 (3126.80) | 19380.8 (5261.89) | 27664.5 (7758.37)

3. Secondary Outcome: PK Parameter: Cmax of Evixapodlin During the Dose Escalation Phase
Description: Cmax was defined as the maximum observed drug concentration.
Time Frame: Intensive PK: Predose, 0.5, 1, 1.5, 2.5, 4, 6, 24 h postdose (400-1500 QD mg cohorts) on C1D1 & D15
Population: Participants in PK Analysis Set were analyzed. Data for Cohort 1 included participants from Cohort 1 and Substudy Cohort 1. PK data were not collected for Cohort 3 Substudy group due to discontinuation of the development program.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Evixapodlin 400 mg (Phase 1) | Cohort 2: Evixapodlin 700 mg (Phase 1) | Cohort 3: Evixapodlin 1000 mg (Phase 1) | Cohort 4: Evixapodlin 1500 mg (Phase 1)
Number analyzed (Participants) | 5 | 3 | 6 | 3
ng/mL
  C1D1 | 1090.4 (355.12) | 1468.7 (497.74) | 1918.3 (377.59) | 2116.7 (55.08)
  C1D15 | 1193.8 (605.87) | 1580.0 (245.76) | 2051.7 (686.89) | 2480.0 (278.75)

4. Secondary Outcome: PK Parameter: Ctrough of Evixapodlin During the Dose Escalation Phase
Description: Ctrough is defined as the observed concentration at the end of the dosing interval.
Time Frame: Intensive PK: Predose, 0.5, 1, 1.5, 2.5, 4, 6, 24 h postdose (400-1500 QD mg cohorts) on C1D1 & D15
Population: Participants in the PK Analysis Set were analyzed. Data for Cohort 1 included participants from Cohort 1 and Substudy Cohort 1. PK data were not collected for Cohort 3 Substudy group due to discontinuation of the development program.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Evixapodlin 400 mg (Phase 1) | Cohort 2: Evixapodlin 700 mg (Phase 1) | Cohort 3: Evixapodlin 1000 mg (Phase 1) | Cohort 4: Evixapodlin 1500 mg (Phase 1)
Number analyzed (Participants) | 5 | 3 | 6 | 3
ng/mL
  C1D1 | 40.3 (9.80) | 56.2 (18.05) | 111.9 (43.92) | 180.3 (21.50)
  C1D15 | 109.8 (35.61) | 198.7 (57.98) | 318.5 (88.44) | 472.7 (112.88)

5. Secondary Outcome: PK Parameter: Tmax of Evixapodlin During the Dose Escalation Phase
Description: Tmax is defined as the time to maximum observed concentration.
Time Frame: Intensive PK: Predose, 0.5, 1, 1.5, 2.5, 4, 6, 24 h postdose (400-1500 QD mg cohorts) on C1D1 & D15
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1: Evixapodlin 400 mg (Phase 1) | Cohort 2: Evixapodlin 700 mg (Phase 1) | Cohort 3: Evixapodlin 1000 mg (Phase 1) | Cohort 4: Evixapodlin 1500 mg (Phase 1)
Number analyzed (Participants) | 5 | 3 | 6 | 3
hours
  C1D1 | 1.00 [1.00 to 1.02] | 1.53 [1.00 to 2.50] | 1.52 [1.00 to 1.65] | 2.50 [2.50 to 6.00]
  C1D15 | 1.50 [1.00 to 2.02] | 1.50 [1.00 to 1.50] | 1.51 [1.00 to 2.50] | 4.00 [1.50 to 5.95]

6. Secondary Outcome: Percentage of Participants Experiencing ≥ Grade 3 Treatment-Emergent Adverse Events During the Dose Expansion Phase
Time Frame: First dose date through end of treatment plus 30 days, approximately 5 years
Population: The study was closed due to sponsor decision prior to opening the dose expansion phase. Hence, no participants were analyzed in this phase.
Groups:
- Dose Expansion (Phase 2): Dose expansion was planned to begin when the recommended Phase 2 dose (RP2D) was determined. The study was closed due to sponsor decision prior to opening the dose expansion cohort and hence RP2D analysis was not performed.
Arm/Group | Dose Expansion (Phase 2)
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants Experiencing ≥ Grade 3 Treatment-Emergent Laboratory Abnormalities During the Dose Expansion Phase
Time Frame: First dose date through end of treatment plus 30 days, approximately 5 years
Population: as for outcome 6
Arm/Group | Dose Expansion (Phase 2)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to 46.1 weeks Adverse Events: First dose date up to last dose (maximum: 39.1 weeks) plus 30 days
Description: All-Cause Mortality: All Enrolled Analysis Set included all participants who received a study identification number in the study after screening.
  Adverse Events: Safety Analysis Set included data from all participants who received at least 1 dose of study treatment, with treatment assignments designated according to the actual treatment received.
Arm/Group | Cohort 1: Evixapodlin 400 mg (Phase 1) | Cohort 2: Evixapodlin 700 mg (Phase 1) | Cohort 3: Evixapodlin 1000 mg (Phase 1) | Cohort 4: Evixapodlin 1500 mg (Phase 1) | Cohort 1 Substudy: Evixapodlin 400 mg (Phase 1) | Cohort 3 Substudy: Evixapodlin 1000 mg (Phase 1)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/3 | 0/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/6 | 1/3 | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3 | 2/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Evixapodlin 400 mg (Phase 1) (N=3) | Cohort 2: Evixapodlin 700 mg (Phase 1) (N=3) | Cohort 3: Evixapodlin 1000 mg (Phase 1) (N=6) | Cohort 4: Evixapodlin 1500 mg (Phase 1) (N=3) | Cohort 1 Substudy: Evixapodlin 400 mg (Phase 1) (N=2) | Cohort 3 Substudy: Evixapodlin 1000 mg (Phase 1) (N=1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Evixapodlin 400 mg (Phase 1) (N=3) | Cohort 2: Evixapodlin 700 mg (Phase 1) (N=3) | Cohort 3: Evixapodlin 1000 mg (Phase 1) (N=6) | Cohort 4: Evixapodlin 1500 mg (Phase 1) (N=3) | Cohort 1 Substudy: Evixapodlin 400 mg (Phase 1) (N=2) | Cohort 3 Substudy: Evixapodlin 1000 mg (Phase 1) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 4 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 4 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to early termination, the study did not proceed to dose expansion phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT04049617/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT04049617/SAP_001.pdf